CLINICAL TRIAL: NCT06508437
Title: Effect of Influenza Vaccination on Global Systemic Inflammatory Markers in Patients With Stable Coronary Artery Disease - Randomized Delayed-Start Pilot Trial
Brief Title: Effect of Influenza Vaccination on Global Systemic Inflammatory Markers in Patients With Stable Coronary Artery Disease
Acronym: IVAMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DR240124
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Inflammatory Response; Atherosclerosis
Keywords: influenza vaccination; inflammation; atherosclerosis,; coronary disease
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Influenza, Human; Inflammation; Coronary Disease | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Immediate" Vaccination Group (Active Comparator): At the inclusion visit (D0), a dose of influenza vaccine will be administered.
  Interventions: Biological: Influenza Vaccination
- "Follow-up" vaccination group (No Intervention): At the inclusion visit (D0), no immediate influenza vaccination (which will be administered one month later at the follow-up visit).

INTERVENTIONS:
Biological: Influenza Vaccination — Standard Dose QIV (15µg Hemagglutinin) - VaxigripTetra Suspension for injection, 0,5ml prefilled syringe
  Arms: "Immediate" Vaccination Group

SUMMARY:
Observational and randomized studies suggest that influenza vaccine may reduce future cardiovascular events in patients with cardiovascular disease. Beyond classical view of indirect effect, linked to the neutralisation of the virus, it is currently considered whether the vaccination may have a direct effect on inflammatory process.Atherosclerosis is known to be driven both by lipid stress and inflammation both at local and systemic level. The investigators suggest that influenza vaccination could have a positive effect on atherosclerosis by regulating plasma inflammation. The aim of this pilot study is therefore to assess the impact of influenza vaccination in patients with stable coronary artery disease on the circulating inflammatory response, in order to validate its potential immunomodulatory effect. If it is found to be beneficial, it could also constitute a future adjuvant therapeutic tool to traditional pharmacotherapy in the prevention of cardiovascular events.

DETAILED DESCRIPTION:
A multi-center, open-label, randomized delayed-start pilot study in 2 parallel groups will be conducted: participants will be randomized as to when the influenza vaccine will be administered, according to a 1:1 ratio between influenza vaccination immediately after inclusion or at 1-month follow-up. Blood tests for plasmatic inflammation analyses will be collected at baseline and at 1 month after study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 60 years.
* With documented stable coronary artery disease.
* Subjects who, in the opinion of the investigator, can comply with the protocol requirements (i.e., show up for the follow-up visit and be able to converse with study staff).
* Signature of free, written and informed consent by the patient.
* Affiliation to a French social security system.

Exclusion Criteria:

* History of serious reaction to influenza vaccine or refusal of vaccination or contraindication to vaccination.
* Participant has received the influenza vaccine within <6 months or another vaccine.
* Acute infection within <3 months or acute worsening of chronic diseases.
* Severe neurocognitive disorders (inability to give informed consent).
* Pre-existing medical conditions or medications involving the immune system (rheumatoid arthritis or other inflammatory conditions or active cancer, recent use (within the past year) of immunosuppressive or modulating agents, including oral steroids, chemotherapy, or radiation therapy) .
* Cardiovascular surgery or other interventions within 6 months preceding the study or planned during the follow-up period.
* Patient's wish or clinical situation requiring co-administration with other vaccines or any factor hindering monitoring.
* Patient under guardianship, curatorship or safeguard of justice.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of high-sensitivity C-reactive protein (hsCRP) | Between baseline and 1-month follow up
  Change from baseline in peripheral blood hsCRP concentrations (mg/L) between study group

SECONDARY OUTCOMES:
Other Plasma inflammatory markers : Tumor necrosis factor alpha (TNF-α), Interleukin 1 beta (IL-1β), Interleukin-6 (IL-6 ) | Between baseline and 1-month follow up
  Change from baseline in peripheral blood markers: Tumor necrosis factor alpha (TNF-α), Interleukin 1 beta (IL-1β), Interleukin-6 (IL-6 ) concentrations (pg/mL) parbetween study group
Other Plasma inflammatory markers : N-terminal pro-B-type natriuretic peptide | Between baseline and 1-month follow up
  Change from baseline in peripheral blood markers N-terminal pro-B-type natriuretic peptide concentrations (ng/L) between study group
Other Plasma inflammatory markers : fibrinogen | Between baseline and 1-month follow up
  Change from baseline in peripheral blood markers: fibrinogen concentrations (g/L) between study group
Plasma arterial vulnerability markers | Between baseline and 1-month follow up
  Change from baseline in peripheral blood markers (g/l) : Apolipoprotein B, lipoprotein(a) and low density lipoproteins cholesterol (LDLc) between study group
Immunoinflammatory markers in circulating immune cells : T cell response | Between baseline and 1-month follow up
  Differences in the expression level of peripheral blood immune cells by reverse transcription and real-time PCR (RT-qPCR) of genes involved in the T-cell response (CD3, CD4, CD8) between study group.
Immunoinflammatory markers in circulating immune cells : T cell population | Between baseline and 1-month follow up
  Differences in the expression level of peripheral blood immune cells by reverse transcription and real-time PCR (RT-qPCR) of genes involved in the T-cell orientation : Th1 (Tbet), Th2 (GATA3), Th17 (RORγ), Treg (FOXP3) between study group.
Circulating immune cells profile : percentage of peripheral immune cells | Between baseline and 1-month follow up
  Differences in peripheral blood immune cells determined by flow cytometry from blood mononuclear cells (PBMC): Percentage of B lymphocytes (CD45+CD19+), T lymphocytes (CD45+CD3+) and monocytes (CD45+CD14+CD11c+) between study group.

CONTACTS AND LOCATIONS:
Locations (1):
- Chru de Trousseau, Tours, France